CLINICAL TRIAL: NCT02225314
Title: Computer-based Cognitive Training for Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADWilliams2012-647173
Record Dates: First submitted 2014-08-19; First posted 2014-08-26 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: Parkinson's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brain Fitness (Experimental): Brain Fitness is a computer-based cognitive training programs designed to augment auditory processing speed and accuracy over an 8-week period to individuals with PD and MCI at a community Parkinson's and Movement Disorders specialty clinic.
  Interventions: Behavioral: Brain Fitness
- InSight (Experimental): InSight is a computer-based cognitive training programs designed to augment visual processing and working memory over an 8-week period to individuals with PD and MCI at a community Parkinson's and Movement Disorders specialty clinic.
  Interventions: Behavioral: InSight
- Active Control (Active Comparator): An active control arm is necessary to model practice effects in an untreated group. Participants in this group will view and complete quizzes on a computerized learning program designed to improve knowledge about literature, art, and history.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Brain Fitness — Brain Fitness is a computer-based cognitive training programs that consists of six types of exercises that train auditory processing speed and accuracy.
  Arms: Brain Fitness
Behavioral: InSight — InSight is a computer-based cognitive training program that consists of five types of exercises that train visual processing and working memory.
  Arms: InSight
Behavioral: Active Control — The Active Control arm is a computerized learning program that consists of five programs (i.e., Wright Brothers, History of Britain, Sister Wendy's American Collection, In Search of Shakespeare, and View the Cosmos) designed to improve knowledge about literature, art, and history.
  Arms: Active Control

SUMMARY:
Computer-Based Cognitive Training for Individuals with Parkinson's Disease" is a 3-arm randomized controlled trial (RCT) comparing Brain Fitness, InSight, and an active control (AC) training program to evaluate the feasibility of empirically supported computer-based cognitive training programs (CCTPs) for patients diagnosed with Parkinson's disease (PD) with Mild Cognitive Impairment (MCI). This pilot study aims to address the need for increased interventions to target non-motor symptoms associated with PD.

DETAILED DESCRIPTION:
Patients meeting criteria for MCI will be initially randomized to one of the 3 conditions. Participants will complete cognitive training exercises on their home or clinic-provided computers for 60 minutes per day, 5 days per week. Compliance and performance will be monitored on a weekly basis and at completion of the study. Outcome measures will be collected one week before initiation of the intervention and within one week completion of the intervention. Neuropsychological functioning, including tests of processing speed, attention, and executive functioning, will serve as primary outcome measures. Patient reported outcomes, including measures of overall QOL and disease-specific QOL, and support-person reported outcomes (if applicable), including measures of overall QOL and caregiver burden, will be secondary outcome measures. This pilot study promises to evaluate computer-based cognitive training in a novel population and expand access to cognitive rehabilitation services, and is designed to improve cognitive functioning and QOL among a wide range of individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study must speak English and have a confirmed medical diagnosis of Parkinson's disease and meet established criteria for MCI in PD (Litvan et al., 2012), defined as individuals with performances of approximately -1 to -2 standard deviations below the mean on at least two tests within five cognitive domains assessed in their clinical neuropsychological evaluations.

Exclusion Criteria:

* Exclusion criteria include diagnosis of PD dementia based on Movement Disorder Society Task Force criteria (Emre et al., 2007) and other PD-associated comorbid conditions (e.g., severe anxiety, depression, excessive daytime sleepiness, or psychosis) that significantly influence cognitive testing (Litvan et al., 2012).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent Accuracy on Cognitive Training Quizzes | Immediate Post-Intervention
  Percent accuracy of cognitive training quizzes from the cognitive training programs of the RCT will be compared. The quizzes are specific to each cognitive training program. The Brain Fitness quiz is comprised of auditory processing and accuracy tasks. The InSight quiz is comprised of visual processing and working memory tasks. The Active Control quiz is comprised of questions about knowledge, literature, art, and history. Due to the differences between the arms with regards to content, the percent accuracy for each participant will be the outcome measure compared across the three study arms.

SECONDARY OUTCOMES:
Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39) | Change from Baseline to 3 Month Follow Up in PDQ-39
  Change in PDQ-39 scores from baseline to 3 month follow up.
California Verbal Learning Test-II Long Delay Free Recall Scaled Score Change Over 3 Months | Change from Baseline in California Verbal Learning Test-II Long Delay Free Recall Scaled Score at 3 Months
  Change from California Verbal Learning Test-II Long Delay Free Recall Scaled Score from Baseline and 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K. Lageman, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Parkinson's and Movement Disorders Center, Richmond, Virginia, United States